CLINICAL TRIAL: NCT02894658
Title: Prospective Fellow Eye Comparison of Traditional Meibomian Gland Disease Treatment Versus a Single Thermal Pulsation Treatment in Patients With Parkinsons Disease
Brief Title: Lipiflow Versus Warm Compresses in Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of equipment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00033387
Record Dates: First submitted 2016-08-29; First posted 2016-09-09 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2022-12

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Lipiflow system (Experimental): Treatment through the use of heat and pulsatile pressure.
  Interventions: Device: LipiFlow system
- Fellow eye warm compresses (Active Comparator): Warm compresses to fellow eye and daily treatment with eyelid scrubs.
  Interventions: Procedure: Warm compresses

INTERVENTIONS:
Device: LipiFlow system — LipiFlow System is an in-office FDA approved treatment that relieves meibomian gland obstruction through the use of heat and pulsatile pressure.
  Arms: Lipiflow system
Procedure: Warm compresses — Warm compresses will be applied to fellow eye and that eye will undergo daily treatment with eyelid scrubs using a warm wash cloth and "no tears" baby shampoo every morning and warm compresses on the eyelids for 5-10 minutes twice a day. Patients will be instructed on how to perform proper lid hygiene at the initial visit.
  Arms: Fellow eye warm compresses

SUMMARY:
The LipiFlow System (TearScience, Morrisville, NC) is an in-office FDA approved treatment for meibomian gland dysfunction. It relieves meibomian gland obstruction through the use of heat and pulsatile pressure. A recent study has observed that a single treatment with the LipiFlow system can decrease dry eye symptoms and objective findings of meibomian gland dysfunction for 1 year. We aim to see if the Lipiflow System will be beneficial in patients with Parkinsons disease who may have difficulty performing normal meibomian gland dysfunction treatment.

DETAILED DESCRIPTION:
Objectives To determine whether a single treatment with thermal pulsation relieves dry eye symptoms (primary objective) and improves objective findings of meibomian gland dysfunction in patients with Parkinsons disease.

Methods and Measures

Design

* Randomized, controlled trial
* Patient eyes will be randomized to either receive a single thermal pulsation treatment the FDA-approved Lipiflow thermal pulsation system or to use traditional eyelid hygiene or to use traditional eyelid hygiene

ELIGIBILITY:
Patients with Parkinsons disease and dry eye attributed to meibomian gland dysfunction

Inclusion Criteria:

* Medical diagnosis of Parkinsons disease
* > 18 years-old
* Reported dry eye symptoms within 3 months of baseline examination with a Standard Patient Evaluation for Eye Dryness (SPEED) score ≥ 6 at baseline visit
* Evidence of meibomian gland obstruction (based on a total meibomian gland secretion score of ≤ 12 for 15 glands of the lower lid)
* Willingness to stop dry eye medications including antibiotics, non-steroidal and anti-inflammatory drugs, and corticosteroids for 2 weeks prior to treatment and during the duration of the study

Exclusion Criteria:

* Active intraocular inflammation
* Ocular surface abnormality that could potentially compromise corneal integrity in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Meibomian gland assessment defined as assessment of 15 glands on the lower eyelid margin using a handheld instrument, the Meibomian Gland Evaluator. | Four visits up to three months
  Expressed secretion characteristics graded on a scale:
  3 (clear liquid secretion)
  2 (cloudy liquid secretion)
  1 (inspissated/toothpaste consistency)
  0 (no secretion)
  Meibomian gland metrics will be calculated:
  A) Total meibomian gland score (sum of the grades for all 15 glands with a range from 0 to 45)
  B) The number of glands secreting any liquid (clear or cloudy liquid with a grade of 2 or 3) of the 15 glands assessed
  C) The number of glands yielding the optimal clear liquid secretion (clear liquid with a grade of 3) of the 15 glands assessed.

SECONDARY OUTCOMES:
Tear break up time | Four visits up to three months
  Tear break up time defined measured with the fluorescein tear break up time (FBUT) method and categorized as follows
  * "Dry" defined as FBUT values of 1-5 seconds
  * "Marginal" defined as FBUT of 6-9 seconds
  * "Normal" defined as FBUT of 10 or greater seconds
Assessment of dry eye symptoms with Ocular Surface Disease Index (OSDI) score before and after treatment | Four visits up to three months
  The OSDI score is assessed on a scale of 0 to 100 with higher scores representing greater disability.
Best spectacle-corrected visual acuity (BSCVA) with high-contrast Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart using the ETDRS-Fast method under standard illumination | Four visits up to three months
Corneal Staining | Four visits up to three months
  • Corneal staining
  * Evaluated with a slit-lamp biomicroscope 90 seconds after instillation of fluorescein dye using a standard strip method
  * Corneal staining is based on the Report of the National Eye Institute/Industry Workshop on Clinical Trials in Dry Eye and will be graded on a scale of 0 (none) - 3 (severe) with a total corneal staining grade range from 0 to 15
SPEED Questionnaire assessment of dry eye symptoms before and after treatment | Four visits up to three months
  SPEED Questionnaire rating of types, frequency, and severity of symptoms. Frequency is grade 0 to 3. Severity is grade 0 to 4. Higher grades represent greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Burden, MD, Principal Investigator — Wake Forest Baptist Health Eye Center

IPD SHARING:
Plan to Share IPD: No